CLINICAL TRIAL: NCT03508167
Title: National, Phase III, Monocentric, Randomized, Double-blind, Controlled, Parallel, to Evaluate the Security and Efficacy of Dorilax® (Fixed Association of Paracetamol 350 mg, Carisoprodol 150 mg and Caffeine 50 mg) Plus Thermal Band Compared to Placebo Plus Thermal Band in the Treatment of Acute Low Back Pain.
Brief Title: Security and Efficacy of Dorilax® (Fixed Association of Paracetamol 350 mg, Carisoprodol 150 mg and Caffeine 50 mg) Plus Thermal Band Compared to Placebo Plus Thermal Band in the Treatment of Acute Low Back Pain.
Acronym: Delfos
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study design will be reformulated
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACH-DRL-03(01/17)
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermal Band plus Dorilax® (Experimental)
  Interventions: Device: Thermal Band; Drug: Dorilax®
- Thermal Band plus Placebo (Other)
  Interventions: Device: Thermal Band; Drug: Placebo

INTERVENTIONS:
Device: Thermal Band — Thermal Band used 8 hours per day
Drug: Dorilax® — 2 tablets, orally. In case of moderate pain, another 2 tablets could be administered, respecting the interval of 8 hours between the administrations.
  Maximum dosage per day: 6 tablets.
  Arms: Thermal Band plus Dorilax®
Drug: Placebo — 2 tablets, orally. In case of moderate pain, another 2 tablets could be administered, respecting the interval of 8 hours between the administrations.
  Maximum dosage per day: 6 tablets.
  Arms: Thermal Band plus Placebo

SUMMARY:
National clinical trial, phase III, monocentric, randomized, double-blind, controlled, parallel, study of superiority, in which two hundred and thirty four (234) participants of both sexes, aged equal or more than 18 years and equal or less than 54 years, will be randomly allocated in one of two treatment groups. The first group will use Dorilax® plus thermal band and the second group will use thermal band plus placebo. The results will show the efficacy and security of Dorilax® and compare the efficiency of Dorilax® and thermal band.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of both sexes aged ≥ (greater than or equal) to 18 years and ≤ (less than or equal) to 54 years;
2. Ability to understand and consent their participation in this clinical study, expressed by signing the Informed Consent Form (ICF);
3. Patient with acute low back pain who responds to the pain period less than or equal to 3 days;
4. Low back pain in intensity Moderate to severe which corresponds to the severity score at least to 2 scores, evaluated by a 6 scores categoric scale;
5. No traumatic low back pain (with no traumatic lesion for at least 7 days before randomization)
6. Low back pain not caused or related to any clinically significant systemic disease, based on investigator evaluation.

Exclusion Criteria:

1. Any finding of clinical observation (clinical / physical assessment) that is interpreted by the investigating physician as a risk to the participation of the research participant in the clinical study;
2. Any laboratorial finding that the Investigator consider a risk to subject of the study;
3. Any finding of a previous imaging examination that the investigator considers to be a risk for clinical study participation;
4. Known hypersensitivity to the components of the medicines used during the study;
5. Women in pregnancy or nursing period;
6. Women who do not agree to use acceptable contraceptive methods (oral contraceptive, intravenous contraceptive, intrauterine device (IUD), hormonal implant, barrier methods, hormonal transdermal patch and tubal ligation); except for those surgically sterile (bilateral oophorectomy or hysterectomy), menopause for at least one year, and participants who report not engaging in sexual practices or non-reproductive practices;
7. Male participants who did not agree to use acceptable methods of contraception;
8. Subjects that has participated in clinical trial protocols in the last twelve (12) months (National Board of Health- Resolution 251 of 07 August 1997, Part III, sub-item J), unless the investigator considers that there may be a direct benefit to it;
9. Subjects who have a relationship of kinship to second degree or any bond with the sponsor or research center employees;
10. Any serious medical illness, at the discretion of the investigator. For example, sciatica that extends below the knee [associated with numbness, tingling, and acute and irradiated pain]) or other neurological deficits (eg, altered straight leg elevation test, abolished or diminished patellar reflex, function of the intestine and / or bladder); Orthopedic surgery history;Fibromyalgia; Diabetes mellitus; peripheral vascular disease; Osteoporosis; Gastrointestinal ulcers; Bleeding or perforation of the gastrointestinal tract; kidney disease; pulmonary edema; Cardiomyopathy; Liver disease; intrinsic defects of coagulation; Hemorrhagic diseases;
11. Any skin lesions (eg rash, bruising, swelling, irritation, laceration, excoriation, ulceration) in the lower back.
12. Use of β-adrenergic blocking agents, antidepressant drugs or supplements that have effects on the central nervous system or that used short- or long-acting analgesic drugs within 24 to 48 hours before randomization, respectively.
13. History of alcohol and / or illicit drug abuse, involvement in active litigation, or worker's compensation claim involving lumbar spine deficiency, back pain for more than 28 consecutive days, or heat hypersensitivity or NSAIDs.
14. Subjects with febrile condition (axillary temperature greater or equal to 37.8ºC)
15. Subjects who have recently had a bacterial infection (last 90 days) that affect the vertebral column, pelvic or abdominal region; as well as participants with a history of bacterial infection that affected the spine in a chronic way;
16. Subjects with unexplained weight loss (more than 10 kg in the last three months);
17. Subjects who are performing some type of oral, physical or topical treatment for low back pain (eg acupuncture, local heat and yoga) and / or initiation of physiotherapy program in the last 2 months before the start of therapy. study;
18. Diabetic subjects, controlled or not.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Compare the efficacy and security of Dorilax® plus thermal banc and Placebo plus thermal band | 8 hours
  The relief of the pain will be evaluated using a 6 points scale.
  0 = no relief; 1 = little relief; 2 = less than half of relief; 3 = more than half of relief; 4 = a lot of relief; 5 = complete relief;
  The first 2 hours will be evaluated at the center and the other 6 hours the subject will need to provide a diary completed hourly with the pain evaluation.

SECONDARY OUTCOMES:
Evaluation of participant satisfaction with treatment | 72 (+24) hours
  Satisfaction of the research participant with the treatment, evaluated in the final visit (VF) by means of the visual analog scale of 100 points (EVA of 100mm, being 0mm = totally unsatisfied and 100mm = totally satisfied).